CLINICAL TRIAL: NCT04176523
Title: Understanding the Long-Term Management of Organic Acidemia Patients With CARBAGLU®: A Mixed Methods Approach
Acronym: PROTECT
Status: Recruiting | Type: Observational
Sponsor: RECORDATI GROUP (Industry)
Responsible Party: Sponsor
Other Study IDs: 17180
Record Dates: First submitted 2019-11-20; First posted 2019-11-25 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Methylmalonic Acidemia; Propionic Acidemia
MeSH Terms: conditions — Methylmalonic acidemia; Propionic Acidemia | interventions — carglumic acid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Methylmalonic_acidemia: Patients with confirmed diagnosis of methylmalonic acidemia, and treated with carglumic acid, at any dose form, any dosage,
  Interventions: Drug: Carglumic Acid
- Propionic_Acidemia: Patients with confirmed diagnosis of propionic acidemia, and treated with carglumic acid, at any dose
  Interventions: Drug: Carglumic Acid

INTERVENTIONS:
Drug: Carglumic Acid — Maintenance therapy with carglumic acid
  Other Names: Carbaglu

SUMMARY:
This is a prospective mixed-design study focused on the long-term management of propionic aciduria (PA) and methylmalonic aciduria (MMA) with N-carbamylglutamate (NCG) maintenance therapy. Treatment characteristics, clinical outcomes, and healthcare utilization data of patients diagnosed PA or MMA treated >6 months therapy with NCG are collected at baseline, 12 months, 18 months, 36 months and 54 months. Qualitative interviews with adult patients and caregivers are conducted >6 months after study enrollment to gain a better understanding of the disease burden and the treatment burden of patients and their families.

DETAILED DESCRIPTION:
Study Design: This is a prospective, longitudinal, observational study of patients diagnosed with organic acidemia that has been on treatment with carglumic acid for a minimum of six months for the long-term management of their disease. This prospective observational study population will include up to 85 diagnosed MMA or PA patients with current carglumic acid treatment experience from 6 European countries: Sweden, the United Kingdom (UK), the Netherlands, Germany, Norway, Italy, Spain and France. The patients (or caregivers) included in this prospective observational study will also be invited to participate in a one-on-one phone interview.

Study Procedures: After Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approval is obtained for the protocol and all supporting protocol documents, clinicians caring for patients with MMA or PA will provide their patients (or caregivers) with the opportunity to participate in the study. Patients (or caregivers) will receive an Information Letter (PIL) (Appendices A and B) inviting them (or their caregiver) to take part in a prospective observational study and in a one-on-one phone interview.

Patients (or caregivers) who are interested in participating in this observational/interview study will review the informed consent form (Appendices C and D) with the clinician and his/her research team. If agreeable, patients (or caregivers) will be asked to sign the consent form and a countersigned copy will be provided to them for their records. Clinicians and their research team at each site will then review patient charts and record demographic and medical history information for each patient. Patient information from medical charts will be collected at the start of the study (baseline), and 12 months and 18 months, and 36 months, and 54 months after baseline. All information derived from medical chart reviews will be recorded through web-based Electronic Data Capture system (EDC).

Patients (or caregivers) who agree to participate in a one-on-one phone interview will provide contact information for their clinicians and the respective research team to include in the Contact Information Form (CIF) (Appendix E). Researchers will then contact patients (or caregivers) directly to schedule a one-hour phone interview. An interview guide (Appendices F and G) including open-ended questions and probes will be used to elicit concepts and orient the discussion during the interview. Patient (or caregiver) interviews will focus on describing the symptoms and impacts of MMA or PA, as well as patient treatment experiences with carglumic acid, their treatment preferences, and their satisfaction with treatment. At the end of the interview, patients (or caregivers) will be asked to complete a Demographic and Health Information Form (DHIF; Appendices H and I). Phone interviews will be audio-recorded with the patient's (or caregiver) permission, transcribed and translated (as needed) in preparation for qualitative analysis.

Data Analysis: The primary prospective data analysis will involve a comparison of the incidence and duration of decompensation episodes pre- and post- initiation of carglumic acid. Additional analysis will include healthcare resource utilization around individual decompensation events, patient/caregiver burden, and patient/caregiver satisfaction with treatment. All prospective data will be undertaken using SAS® software, version 9.4 of the SAS® system for Windows (Cary, NC, USA). All qualitative data from the interviews will be analyzed using ATLAS.ti, a software package uniquely designed to analyze qualitative data. The audio-recorded verbatim transcripts of the interviews will be coded to identify patterns in participants' responses concerning patient experiences with the symptoms and impacts of MMA or PA, treatment experience with carglumic acid, patient treatment preferences, and treatment satisfaction. Findings will be summarized in a final report and may be published or presented by the investigator(s) after the review by, and in consultation and agreement with, the sponsor. If published or presented, the results will be presented in such a way that confidential or proprietary information is not disclosed.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has confirmed diagnosis of an organic acidemia (e.g., MMA or PA)
2. Patient initiated treatment with carglumic acid for long-term management of MMA or PA
3. Patient has been treated with carglumic acid for a minimum of 6 months
4. Patient (or caregiver) is able to comply with all prospective study procedures
5. Patient (or caregiver) is able to provide informed consent

Exclusion Criteria:

* None

Ages: 6 Months to 99 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with organic acideamia that have been on treatment with CARBAGLU® for a minimum of six months for the long-term management of their disease. This prospective observational study population will include up to 95 diagnosed MMA or PA patients with current carglumic acid treatment experience from 6 European countries: Sweden, the United Kingdom (UK), the Netherlands, Germany, Norway, Italy, Spain and France. The patients (or caregivers) included in this prospective observational study will also be invited to participate in a one-on-one phone interview.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Estimated)
Dates: Start 2019-01-15 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2029-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in Number and Duration of Decompensation Events | 54 months
  Change in the number of decompensation events before and after treatment with carglumic acid

SECONDARY OUTCOMES:
Frequency and Duration of Healthcare Resource Utilization | 18 months
  Estimation of the health care resource utilization associated with a decompensation event with number of inpatient hospitalization vs. outpatient vs. home. Treatment used to control ammonia levels during decompensation episodes. Number of emergency visits. number of visits to specialist or to general practitioner. Number of hospital stays. Number of bed days in hospital.
Caregiver Burden Exposure Frequency and Duration | 18 months
  description of the patient and caregiver burden associated with MMA and PA
Caregiver Satisfaction Level | 18 months
  Describe the MMA and PA patient and caregiver satisfaction with MMA or PA treatment
Maintenance Dosage of NCG | 54 months
  Document the dosages of NCG used in maintenance treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sufin Yap, MD, Principal Investigator — Sheffield Children's NHS Trust
Locations (32):
- France (8):
  - Hopital Des Enfants, CHU de Bordeaux-GH Pellegrin, Bordeaux
  - Hopital de la Conception, Marseille
  - Hôpital de la Timone, Marseille
  - CHU de Nancy - Hopitaux de Brabois, Nancy
  - Hôpital Necker Enfants Malades, Paris
  - CHU de Rouen, Rouen
  - Nouvel Hopital Civil, Strasbourg
  - Hopital de Hautepierre, Strasbourg
- Klinikum Bremen Mitte, Prof. Hess Kinderklinik, Bremen, Germany
- Italy (7):
  - Azienda Ospedaliero Universitaria Meyer, Florence
  - San Paola Hospital, ASST Santi Paolo e Carlo, Milan
  - Milan Policlinico University, Milan
  - Azienda Ospedaliera San Gerardo Monza, Monza
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - University Hospital of Padova, Padua
  - Turin University Hospital, Turin
- Oslo University Hospital, Oslo, Norway
- Spain (11):
  - AMM hospital val d'hebron, Barcelona
  - Sant Joan de Deu, Barcelona
  - Universitario de Cruces, Bilbao
  - Hospital Infantil Universitario Nino Jesus, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Universitario Ramon y Cajal Madrid, Madrid
  - Hospital Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitario Son Espases, Palma de Mallorca
  - Hospital Universitario Virgen del Rocio, Seville
  - Universitario Miguel Servet, Zaragoza
- NÄL, Trollhättan, Sweden
- United Kingdom (3):
  - Guy's and St. Thomas' Hospital NHS Foundation Trust, London
  - Great Ormond Street Hospital, London
  - Sheffield Children's Hospital NHS Foundation Trust, Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burlina A, Bettocchi I, Biasucci G, Bordugo A, Gasperini S, La Spina L, Maines E, Meli C, Menni F, Paci S, Procopio E, Rossi A, Rubert L, Spada M, Tubili F, Tummolo A. Long-term use of carglumic acid in methylmalonic aciduria, propionic aciduria and isovaleric aciduria in Italy: a qualitative survey. Eur Rev Med Pharmacol Sci. 2022 Jul;26(14):5136-5143. doi: 10.26355/eurrev_202207_29302. PMID 35916811
- [Background] Alfadhel M, Nashabat M, Saleh M, Elamin M, Alfares A, Al Othaim A, Umair M, Ahmed H, Ababneh F, Al Mutairi F, Eyaid W, Alswaid A, Alohali L, Faqeih E, Almannai M, Aljeraisy M, Albdah B, Hussein MA, Rahbeeni Z, Alasmari A. Long-term effectiveness of carglumic acid in patients with propionic acidemia (PA) and methylmalonic acidemia (MMA): a randomized clinical trial. Orphanet J Rare Dis. 2021 Oct 11;16(1):422. doi: 10.1186/s13023-021-02032-8. PMID 34635114
- [Background] Kido J, Matsumoto S, Nakamura K. Carglumic Acid Contributes to a Favorable Clinical Course in a Case of Severe Propionic Acidemia. Case Rep Pediatr. 2020 Mar 9;2020:4709548. doi: 10.1155/2020/4709548. eCollection 2020. PMID 32231837
- [Background] Kiykim E, Oguz O, Duman C, Zubarioglu T, Cansever MS, Zeybek ACA. Long-term N-carbamylglutamate treatment of hyperammonemia in patients with classic organic acidemias. Mol Genet Metab Rep. 2021 Jan 30;26:100715. doi: 10.1016/j.ymgmr.2021.100715. eCollection 2021 Mar. PMID 33552909
- [Background] Tummolo A, Melpignano L, Carella A, Di Mauro AM, Piccinno E, Vendemiale M, Ortolani F, Fedele S, Masciopinto M, Papadia F. Long-term continuous N-carbamylglutamate treatment in frequently decompensated propionic acidemia: a case report. J Med Case Rep. 2018 Apr 22;12(1):103. doi: 10.1186/s13256-018-1631-1. PMID 29679984
- [Background] Burlina A, Cazzorla C, Zanonato E, Viggiano E, Fasan I, Polo G. Clinical experience with N-carbamylglutamate in a single-centre cohort of patients with propionic and methylmalonic aciduria. Mol Genet Metab Rep. 2016 Jul 13;8:34-40. doi: 10.1016/j.ymgmr.2016.06.007. eCollection 2016 Sep. PMID 27489777
- [Background] Yap S, Lamireau D, Feillet F, Ruiz Gomez A, Davison J, Tangeraas T, Giordano V. Real-World Experience of Carglumic Acid for Methylmalonic and Propionic Acidurias: An Interim Analysis of the Multicentre Observational PROTECT Study. Drugs R D. 2024 Mar;24(1):69-80. doi: 10.1007/s40268-023-00449-z. Epub 2024 Jan 10. PMID 38198106